CLINICAL TRIAL: NCT03201952
Title: Examination of the Metabolic Effects of Direct Bile Salt Delivery to the Ileum in Humans
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty in participant recruitment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Dole, Clinical Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 162023
Record Dates: First submitted 2017-06-22; First posted 2017-06-28 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Glucose Intolerance; Gastric Bypass Surgery
Keywords: Glucose; Ileostomy
MeSH Terms: conditions — Glucose Intolerance | interventions — Ursodeoxycholic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Each volunteering subject will participate in 2 study visits, receiving the placebo at one visit and investigation medication at the other visit. The order of these visits will be randomized.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ursodeoxycholic Acid/Placebos (Active Comparator): During one of the subjects two randomized visits the subject will receive a 300mg elixir solution of ursodeoxycholic acid (UDCA) via their ileostomy that has been prepared by investigational drug services (IDS) in a 5cc elixir formulation during visit #1. During visit #2 subjects will receive a saline solution of totaling 5cc via their ileostomy that has been prepared by investigational drug services (IDS) in order to mimic the preparation of the medication comparator of ursodeoxycholic acid.
  Interventions: Drug: Ursodeoxycholic Acid; Drug: Placebos
- Placebos/Ursodeoxycholic Acid (Active Comparator): Subjects will receive a saline solution of totaling 5cc via their ileostomy that has been prepared by investigational drug services (IDS) in order to mimic the preparation of the medication comparator of ursodeoxycholic acid during visit #1. During visit #2 subject will receive a 300mg elixir solution of ursodeoxycholic acid (UDCA) via their ileostomy that has been prepared by investigational drug services (IDS) in a 5cc elixir formulation.
  Interventions: Drug: Ursodeoxycholic Acid; Drug: Placebos

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — Ileostomy administration of 300mg UDCA once
  Other Names: UDCA
Drug: Placebos — Ileostomy administration of 5cc saline placebo once
  Other Names: Saline

SUMMARY:
This project will evaluate distal intestinal bile salt administration in humans by deliving ursodeoxycholic acid (UDCA) into the terminal ileum of subjects with a pre-existing ileostomy and assessing several hormone levels following an oral glucose tolerance test compared to a placebo.

DETAILED DESCRIPTION:
Ursodeoxycholic acid (UDCA) is currently FDA-approved for the treatment of gallstone dissolution and primary biliary cirrhosis. Other than these two diseases, exploratory research - both preclinical and clinical - has demonstrated other beneficial effects of UDCA. For example, systemic administration of UDCA for several weeks (4-6 weeks) has been shown to improve insulin sensitivity in non-diabetic, obese individuals. Whether or not these effects on insulin sensitivity may be acute in nature and are detectable by OGTT are unknown. Based on growing knowledge of bile salt receptors in the gastrointestinal tract, at least some of these effects of bile salts on metabolism appear to be mediated by receptors constitutively expressed in the terminal ileum (e.g. TGR5 receptor that is upstream of GLP-1 and insulin secretion that control blood glucose levels). Thus, metabolic effects may be inducible with acute UDCA administration directly into this region of the intestine that could be useful in screening compounds or designing future mechanistic studies. This pilot study is designed to examine the effects of UDCA on oral glucose tolerance versus a placebo in non-diabetic across a range of body mass indexes by infusing UDCA directly into the ileum of volunteering subjects with a pre-existing ileostomy and measuring hormone response. The investigators aim to recruit approximately 4-5 volunteers in a lean BMI range (18.5-25 kg/m2), overweight (>25-29.9), class 1 obesity (>30-35 kg/m2), and class 2 obesity (>35-40 kg/m2) for a total of ~16-20 participants.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Presence of an ileostomy > 2 months
* Weight stable* for >2 months (i.e. no greater than 7% change in body weight the last 2 months)

Exclusion Criteria:

* Crohn's Disease
* Steroid use in the last 3 months
* Documented/known diagnosis of type 1 diabetes or type 2 diabetes, chronic liver disease, chronic kidney disease, heart failure, cardiac dysrhythmias, or familial hypercholesterolemia
* Current use of any over-the-counter or prescription oral bile salt
* Currently pregnant
* Current use of medications that are known to interact with Ursodiol
* Current or former smoker within the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in glucose level | 3 hours
  Following UDCA administration and a 2 hour period to allow steady state, a 3 hour glucose tolerance test will be completed while measuring glucose change from baseline.

SECONDARY OUTCOMES:
Change in insulin Level | Baseline to 3 hours
  Following UDCA administration and a 2 hour period to allow steady state, a 3 hour glucose tolerance test will be completed while measuring insulin level
Change in GLP-1 Level | Baseline to 3 hours
  Following UDCA administration and a 2 hour period to allow steady state, a 3 hour glucose tolerance test will be completed while measuring GLP-1

CONTACTS AND LOCATIONS:
Overall Officials: Naji Abumrad, MD, Study Director — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Albaugh VL, Flynn CR, Cai S, Xiao Y, Tamboli RA, Abumrad NN. Early Increases in Bile Acids Post Roux-en-Y Gastric Bypass Are Driven by Insulin-Sensitizing, Secondary Bile Acids. J Clin Endocrinol Metab. 2015 Sep;100(9):E1225-33. doi: 10.1210/jc.2015-2467. Epub 2015 Jul 21. PMID 26196952
- [Background] Flynn CR, Albaugh VL, Cai S, Cheung-Flynn J, Williams PE, Brucker RM, Bordenstein SR, Guo Y, Wasserman DH, Abumrad NN. Bile diversion to the distal small intestine has comparable metabolic benefits to bariatric surgery. Nat Commun. 2015 Jul 21;6:7715. doi: 10.1038/ncomms8715. PMID 26197299